CLINICAL TRIAL: NCT02394899
Title: Integrating a Parenting Intervention With Routine Care to Improve Parental Psychosocial Functioning and Early Developmental Outcomes in Children With Sickle Cell Disease
Brief Title: Improving Parental Psychosocial Functioning and Early Developmental Outcomes in Children With Sickle Cell Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of The West Indies (Other)
Collaborators: Grand Challenges Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0001
Record Dates: First submitted 2015-02-04; First posted 2015-03-20 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Sickle Cell Disease; Cognitive Ability, General; Psychological Stress; Parenting
Keywords: SCD; early childhood intervention; parental stress; neurocognition
MeSH Terms: conditions — Anemia, Sickle Cell; Stress, Psychological | interventions — Play Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): The control dyad will receive usual care.
- Intervened (Experimental): Parents receive training in problem solving skills and play therapy with their infants.
  Interventions: Behavioral: Play therapy; Other: Problem solving skills

INTERVENTIONS:
Behavioral: Play therapy — Short films that have been developed to deliver a series of child development messages will be shown at the monthly visits. Nine modules of approximate length 3 minutes each have been developed and cover the topics: Love, Comforting baby, Talking to babies and children, Praise, Using bath time to play and learn, Looking at books, Simple toys mothers can make, Drawing and games, and Puzzles. Nurses at the Sickle cell Unit (SCU) will be trained to discuss the video messages with the mothers/caregivers, demonstrate activities they can do with their children and how to make simple toys from household materials. Mothers/caregivers will practice some of the activities and they will be encouraged to make them part of their daily routine.
  Arms: Intervened
Other: Problem solving skills — Problem solving therapy (PST) aims to empower patients or caregivers in attending to daily challenges. It is based on cognitive behavioural therapy and can be used in primary care settings. It encourages persons to use existing resources and skills to function better and find solutions to problems. It will be delivered in 6 sessions over the 6-week period and will last for about 30 minutes per session. The stages of PST are: identification of the problems; generating possible solutions; evaluating and implementing preferred solution; and evaluating to see if the solutions were successful. The parent/caregiver will be taught a process of problem solving with reference to general everyday problems as well as specific problems which may arise while parenting a child with SCD.
  Arms: Intervened

SUMMARY:
There are all significant risk factors for poor early cognitive development and, as such, neurocognitive deficits have been demonstrated in pre-school children with sickle cell disease (SCD). This project assesses the efficacy of using an evidence-based early stimulation program, combined with components to help parents cope with stress, delivered during six routine monthly clinic visits to parents of children with sickle cell disease. It is hoped that this innovation will improve parental psychological outcomes, as well as child developmental outcomes.

DETAILED DESCRIPTION:
Children with sickle cell disease (SCD) are at risk of various complications, many of which arise suddenly and call on the problem solving skills of their parents. They are also at risk of neurocognitive delays; these may become evident during the pre-school years. Previous research by this group has demonstrated improved developmental outcomes after parental interventions incorporating play techniques in high risk and healthy pre-school children. The aim of the study is to determine usefulness in children with SCD of similar developmental interventions augmented by lessons in problem solving.

The study is a randomized controlled trial. Parents of all infants with Hb SS (homozygous sickle cell disease) or Sβ0 -thalassemia disease identified by newborn screening during the initial year of the study will be invited to participate. They will be randomized to intervention or control. Parental stress, infant's development and hemoglobin levels will be measured at recruitment and again after six months. The intervention will occur during monthly Penadur (intramuscular Benzathine Penicillin) visits and will include supervised play with their children using an inexpensive toy and participation in solving a problem which may arise as they parent their child with SCD. At the end of the study, all control dyads will also be given the toys used in the intervention. All parents will be given the results of their children's developmental assessments and appropriate referrals made if deficits are identified.

The study is minimal risk. Every effort will be made to maintain patient confidentiality. Respect for, and the maximum protection of the best interests of the research subjects will be maintained.

ELIGIBILITY:
Inclusion Criteria:

* Infant has sickle cell disease: SS or Sβ0 thalassemia
* Attending Sickle Cell Unit, Jamaica for routine care

Exclusion Criteria:

* None

Ages: 6 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2014-10; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Infant's development quotient (Griffiths Developmental Scale) | 6 months
  Griffiths Developmental Scale
Parental stress, depression and coping (Pediatric Inventory for Parents; CES-D; Coping Health Inventory for parents) | 6 months
  Questionnaires to assess: Pediatric Inventory for Parents; CES-D; Coping Health Inventory for parents
Parental problem solving skills (Social Problem Solving Inventory) | 6 months
  Using Social Problem Solving Inventory: Questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Knight-Madden, MBBS, PhD, Principal Investigator — The University of The West Indies
Locations (1):
- Sickle Cell Unit, University of West Indies, Mona Campus, Kingston, Jamaica